CLINICAL TRIAL: NCT07355036
Title: The Effect of Basic Life Support Training Given by the Escape Room Method on the Knowledge and Skills of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Gülcan Dürüst Sakallı, Dr. lecturer, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EasternMU-SBF-HB-GDS-03
Record Dates: First submitted 2025-04-28; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Education; Nursing Students; Cardio Pulmonary Resuscitation; Nursing Students Education on Cardio Pulmonary Resuscitation; Escape Room
Keywords: escape room; nursing students education; cardio pulmonary resuscitation; basic life support

STUDY DESIGN:
Intervention Model Description: Data collection will begin after ethics committee and institutional permission. All students who accept the study will be randomly assigned to the game and control groups using Random Allocation Software (Random Alloc, Ver. 2.0.0) and the data collection process will be completed. In this study, the game will be applied to the students in the game group by providing escape room training method and basic life support application training. Before the game process, the game scenario will be explained in detail to the students in the intervention groups. The students in the control group will be evaluated by practicing with a CPR simulator. All forms will be applied to the students in both groups.
  Unlike the control group, the students in the intervention groups will be asked to fill out the "Game Evaluation Form". All students will receive the same theoretical training, but the effect of the training model on their knowledge and skills will be evaluated by using different training method
Who Masked: Participant, Care Provider
Masking Description: Data collection will begin after ethics committee and institutional permission. All students who accept the study will be randomly assigned to the game and control groups using Random Allocation Software (Random Alloc, Ver. 2.0.0) and the data collection process will be completed. In this study, the game will be applied to the students in the game group by providing escape room training method and basic life support application training. Before the game process, the game scenario will be explained in detail to the students in the intervention groups. The students in the control group will be evaluated by practicing with a CPR simulator. All forms will be applied to the students in both groups.
  Unlike the control group, the students in the intervention groups will be asked to fill out the "Game Evaluation Form". All students will receive the same theoretical training, but the effect of the training model on their knowledge and skills will be evaluated by using different training method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- escape room group (Experimental): In this study, the game will be applied to the students in the game group by giving basic life support application training with escape room training method. Before the game process, the game scenario will be explained in detail to the students in the game group.
  With randomization, students assigned to the escape room group will carry out the activity using a game prepared with a scenario designed by researchers and evaluated by experts in the field. During the activity, researchers will observe and assess the data using a skill form. The completion times for the activity will be recorded. The pre-test knowledge test, the post-test knowledge test, and the knowledge test taken one month later will be compared.
  Interventions: Other: Experimental escape room group; Other: plasebo control group
- control group (Placebo Comparator): Students in the control group will be evaluated by practicing with a CPR simulator. With randomization, students assigned to the placebo (control) group in this group will perform the procedure using the standard BASIC LIFE SUPPORT (ADULT) SIMULATOR MANIKIN by the researchers. During the procedure, the researchers will observe and evaluate the data using a skills form. The pre-test knowledge test, the post-test knowledge test, and the knowledge test taken one month later will be compared.
  Interventions: Other: Experimental escape room group; Other: plasebo control group

INTERVENTIONS:
Other: Experimental escape room group — With randomization, students assigned to the escape room group will carry out the activity using a game prepared with a scenario designed by researchers and evaluated by experts in the field. During the activity, researchers will observe and assess the data using a skill form. The completion times for the activity will be recorded. The pre-test knowledge test, the post-test knowledge test, and the knowledge test taken one month later will be compared.
Other: plasebo control group — With randomization, students assigned to the placebo (control) group in this group will perform the procedure using the standard BASIC LIFE SUPPORT (ADULT) SIMULATOR MANIKIN by the researchers. During the procedure, the researchers will observe and evaluate the data using a skills form. The pre-test knowledge test, the post-test knowledge test, and the knowledge test taken one month later will be compared.

SUMMARY:
Today, nursing education is not only about the transfer of theoretical information, but also includes the acquisition of multidimensional skills such as clinical decision making, critical thinking and teamwork. In this context, educational escape room games stand out as an effective teaching strategy, especially in basic life support (BLS) applications that require emergency management (Adams, Burger, Crawford & Setter, 2018; Gómez-Urquiza et al., 2019).

Escape room games are team-based, interactive and gamified learning environments in which participants solve puzzles by cooperating within a certain scenario in a limited time and try to achieve the specified goal (Nicholson, 2015; Wiemker, Elumir & Clare, 2015; Clarke et al., 2017). In the teaching of emergency interventions such as cpr, which require time management, quick decision making and coordinated teamwork, this game structure enables students to develop both knowledge and skills (Tassemeyer, Glover & Steve

ELIGIBILITY:
Inclusion Criteria:

Criteria for inclusion in the sample;

* Being older than 18 years of age
* Being a 4th grade student in the Department of Nursing Turkish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Measurement of Adult Basic Life Support Application Knowledge | This evaluation will be conducted before the application, immediately after the application, and again one week later.
  0-50 points is bad, 50-80 points is average, 80-100 points is good.

SECONDARY OUTCOMES:
Measurement of Self-Efficacy of Basic Resuscitation Skills | The Self-Efficacy Measurement for Basic Resuscitation Skills will be administered on the day of the training and again 1 month after the training.
  as the score increases, it shows that his skill is good

OTHER OUTCOMES:
Measurement of Basic Resuscitation Skills Self-Efficacy | This evaluation form will be administered on the day of the intervention and will also be repeated one month after the intervention.
  The score definition here is that the student assigns themselves a score between 0 and 100; each question relates to their self-efficacy regarding the subject. As the score increases, the student considers themselves sufficiently competent in the subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University Cyprus, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33896925/